CLINICAL TRIAL: NCT07400432
Title: Acute Effects of Moderate-Intensity Continuous Exercise Versus High-Intensity Interval Training on Cognitive Performance and Psychophysiological Responses in Physically Active Adults: A Randomized Crossover Study
Brief Title: Acute Effects of Moderate-Intensity Continuous Exercise Versus HIIT on Cognitive Performance and Psychophysiological Responses in Physically Active Adults
Acronym: EXCOG
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Maged Basha, Associate Professor, Consultant, Physical therapy and rehabilitation, Qassim University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: QU 10-20-26
Record Dates: First submitted 2026-01-30; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Sustained Attention; Cognitive Performance; Cognitive Performance During Physical Activity
Keywords: Exercise; High-Intensity Interval Training; Aerobic Exercise; SART; Psychomotor Vigilance Task; Exercise Intensity
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: This study uses a randomized within-subject crossover design in which each participant completes two exercise interventions-moderate-intensity continuous exercise and high-intensity interval training-on separate days, with a 48-72-hour washout period. The order of the interventions is randomized so that each participant serves as their own control.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the exercise interventions, participant and care provider blinding is not feasible. However, cognitive outcome assessors are blinded to the intervention order to minimize assessment bias. Data analysis will be performed using coded datasets to ensure objectivity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate-Intensity Continuous Exercise (MICE) (Experimental): Participants perform continuous treadmill exercise for 20 minutes at 60-70% of age-predicted maximum heart rate, including standardized warm-up and cool-down periods. Heart rate, oxygen saturation, and perceived exertion are monitored throughout the session to ensure protocol adherence and participant safety.
  Interventions: Other: Moderate-Intensity Continuous Exercise (MICE)
- High-Intensity Interval Training (HIIT) (Experimental): Participants perform treadmill-based high-intensity interval training consisting of repeated short bouts at 85-95% of age-predicted maximum heart rate interspersed with brief recovery periods, with a total session duration of approximately 20 minutes including warm-up and cool-down. Heart rate, oxygen saturation, and perceived exertion are continuously monitored.
  Interventions: Other: High-Intensity Interval Training (HIIT)

INTERVENTIONS:
Other: Moderate-Intensity Continuous Exercise (MICE) — Participants perform continuous treadmill exercise for 20 minutes at 60-70% of age-predicted maximum heart rate. Each session includes a standardized warm-up period of approximately 3 minutes and a cool-down period of 2-3 minutes. Heart rate, oxygen saturation, and rating of perceived exertion are monitored throughout the session to ensure adherence to the target intensity and participant safety.
  Other Names: Moderate Aerobic Exercise; Continuous Aerobic Exercise
  Arms: Moderate-Intensity Continuous Exercise (MICE)
Other: High-Intensity Interval Training (HIIT) — Participants perform treadmill-based high-intensity interval training consisting of repeated short bouts of exercise at 85-95% of age-predicted maximum heart rate, interspersed with brief recovery periods. Total session duration is approximately 20 minutes, including standardized warm-up and cool-down periods. Heart rate, oxygen saturation, and rating of perceived exertion are continuously monitored to ensure safety and protocol compliance.
  Other Names: High-Intensity Interval Exercise; Interval Aerobic Training
  Arms: High-Intensity Interval Training (HIIT)

SUMMARY:
This study aims to compare the immediate effects of two common types of exercise-moderate-intensity continuous exercise and high-intensity interval training (HIIT)-on attention, alertness, and physiological responses in physically active young adults.

Attention and mental alertness are essential for learning, academic performance, and daily functioning. Previous research suggests that a single session of exercise can temporarily improve cognitive performance, but it is not clear whether moderate exercise or high-intensity interval exercise is more effective in producing these immediate benefits.

In this study, participants will complete two supervised treadmill exercise sessions on separate days: one session of moderate-intensity continuous exercise and one session of high-intensity interval training. The order of the two exercise sessions will be randomized, and there will be a rest period of 48 to 72 hours between sessions.

Before and immediately after each exercise session, participants will complete computerized cognitive tests that measure sustained attention and reaction time. Heart rate, oxygen saturation, perceived exertion, mood, and alertness will also be measured to evaluate physiological and psychological responses to exercise.

By comparing the effects of these two exercise approaches within the same individuals, this study aims to identify which type of exercise leads to better immediate cognitive performance and favorable physiological responses. The findings may help guide exercise recommendations for improving attention, alertness, and overall mental performance in young adults.

DETAILED DESCRIPTION:
This study is a randomized within-subject crossover clinical trial designed to compare the acute effects of moderate-intensity continuous exercise (MICE) and high-intensity interval training (HIIT) on cognitive performance and psychophysiological responses in physically active young adults.

Each participant will complete two supervised treadmill exercise sessions-one MICE session and one HIIT session-on separate days, with a 48-72-hour washout period. The order of the two exercise conditions will be randomized using a computer-generated sequence. This crossover design allows each participant to serve as their own control, reducing inter-individual variability and increasing statistical power.

Cognitive performance will be assessed immediately before and after each exercise session using validated computerized tests of sustained attention and vigilance, including the Sustained Attention to Response Task (SART) and the Psychomotor Vigilance Task (PVT). Primary cognitive outcomes will include reaction time, accuracy, response inhibition, and attentional lapses.

Psychophysiological responses will be monitored throughout the exercise sessions and immediately post-exercise. These include heart rate, oxygen saturation, rating of perceived exertion, mood, and alertness. Exercise intensity will be prescribed based on percentages of age-predicted maximum heart rate and continuously monitored to ensure protocol adherence and participant safety.

Data will be analyzed using within-subject statistical comparisons to evaluate differences between exercise conditions. The findings are expected to provide evidence on how acute exercise intensity influences immediate cognitive and physiological responses, informing exercise recommendations for optimizing attention and alertness in young adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 30 years.
* Physically active individuals, as assessed by the International Physical Activity Questionnaire (IPAQ).
* In good general health.
* Cleared for physical activity participation based on the Physical Activity Readiness Questionnaire (PAR-Q).
* Enrolled as university students.
* Able and willing to provide written informed consent.

Exclusion Criteria:

* History of cardiovascular, neurological, or musculoskeletal disorders that may affect exercise safety or cognitive performance.
* Presence of uncontrolled hypertension, recent concussion, or any medical condition contraindicating exercise.
* Use of medications that may influence cognition, mood, or cardiovascular responses.
* Pregnancy.
* Failure to pass PAR-Q screening without medical clearance.
* Heavy smoking or history of substance abuse.
* Visual or hearing impairments that could interfere with computerized cognitive task performance.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
Sustained Attention to Response Task (SART) Performance | Immediately before each exercise session (within the same day for both intervention conditions)
  Sustained attention and response inhibition will be assessed using the Sustained Attention to Response Task (SART). Outcome variables will include reaction time, accuracy, commission errors, and omission errors, reflecting participants' ability to maintain sustained attention and inhibitory control following acute exercise.
Sustained Attention to Response Task (SART) Performance | immediately after each exercise session (within the same day for both intervention conditions)
  Sustained attention and response inhibition will be assessed using the Sustained Attention to Response Task (SART). Outcome variables will include reaction time, accuracy, commission errors, and omission errors, reflecting participants' ability to maintain sustained attention and inhibitory control following acute exercise.
Psychomotor Vigilance Task (PVT) Performance | Immediately before each exercise session (within the same day for both intervention conditions)
  Vigilance and reaction time will be evaluated using the Psychomotor Vigilance Task (PVT). Outcome variables will include mean reaction time, number of attentional lapses, and response accuracy, reflecting participants' sustained alertness following acute exercise.
Psychomotor Vigilance Task (PVT) Performance | immediately after each exercise session (within the same day for both intervention conditions)
  Vigilance and reaction time will be evaluated using the Psychomotor Vigilance Task (PVT). Outcome variables will include mean reaction time, number of attentional lapses, and response accuracy, reflecting participants' sustained alertness following acute exercise.

SECONDARY OUTCOMES:
Heart Rate Response During and After Exercise | During each exercise session
  Heart rate will be continuously monitored during each exercise session and recorded at baseline, during exercise, and immediately post-exercise to evaluate physiological responses to moderate-intensity continuous exercise and high-intensity interval training.
Heart Rate Response During and After Exercise | Immediately after each exercise session
  Heart rate will be continuously monitored during each exercise session and recorded at baseline, during exercise, and immediately post-exercise to evaluate physiological responses to moderate-intensity continuous exercise and high-intensity interval training.
Oxygen Saturation (SpO₂) Response | During each exercise session
  Peripheral oxygen saturation will be measured using a pulse oximeter before, during, and immediately after each exercise session to assess acute cardiorespiratory responses to exercise intensity.
Oxygen Saturation (SpO₂) Response | Immediately after each exercise session
  Peripheral oxygen saturation will be measured using a pulse oximeter before, during, and immediately after each exercise session to assess acute cardiorespiratory responses to exercise intensity.
Rating of Perceived Exertion Assessed by the Borg Rating of Perceived Exertion Scale (6-20) | During each exercise session
  Perceived exertion will be assessed using the Borg Rating of Perceived Exertion (RPE) Scale (6-20) during and immediately after each exercise session to evaluate subjective exercise intensity and effort. The scale ranges from 6 (no exertion at all) to 20 (maximal exertion). Higher scores indicate greater perceived physical effort.
Rating of Perceived Exertion Assessed by the Borg Rating of Perceived Exertion Scale (6-20) | Immediately after each exercise session
  Perceived exertion will be assessed using the Borg Rating of Perceived Exertion (RPE) Scale (6-20) during and immediately after each exercise session to evaluate subjective exercise intensity and effort. The scale ranges from 6 (no exertion at all) to 20 (maximal exertion). Higher scores indicate greater perceived physical effort.
Mood and Alertness Assessed by Numeric Rating Scales (0-10) | Immediately before each exercise session
  Subjective mood and alertness will be assessed using separate 10-point Numeric Rating Scales (0-10) administered immediately before and immediately after each exercise session. For each scale, 0 represents the lowest level (very poor mood / extremely sleepy) and 10 represents the highest level (excellent mood / fully alert). Higher scores indicate better mood and greater alertness.
Mood and Alertness Assessed by Numeric Rating Scales (0-10) | Immediately after each exercise session
  Subjective mood and alertness will be assessed using separate 10-point Numeric Rating Scales (0-10) administered immediately before and immediately after each exercise session. For each scale, 0 represents the lowest level (very poor mood / extremely sleepy) and 10 represents the highest level (excellent mood / fully alert). Higher scores indicate better mood and greater alertness.

CONTACTS AND LOCATIONS:
Locations (1):
- Qassim University, Buraidah, Al-Qassim Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly. All collected data will be analyzed and reported in aggregate form only to ensure participant confidentiality and data protection.

REFERENCES:
- [Background] Nanda B, Balde J, Manjunatha S. The Acute Effects of a Single Bout of Moderate-intensity Aerobic Exercise on Cognitive Functions in Healthy Adult Males. J Clin Diagn Res. 2013 Sep;7(9):1883-5. doi: 10.7860/JCDR/2013/5855.3341. Epub 2013 Sep 10. PMID 24179888
- [Background] Pujari V. Moving to Improve Mental Health - The Role of Exercise in Cognitive Function: A Narrative Review. J Pharm Bioallied Sci. 2024 Feb;16(Suppl 1):S26-S30. doi: 10.4103/jpbs.jpbs_614_23. Epub 2024 Feb 29. PMID 38595617
- [Background] Singh B, Bennett H, Miatke A, Dumuid D, Curtis R, Ferguson T, Brinsley J, Szeto K, Petersen JM, Gough C, Eglitis E, Simpson CE, Ekegren CL, Smith AE, Erickson KI, Maher C. Effectiveness of exercise for improving cognition, memory and executive function: a systematic umbrella review and meta-meta-analysis. Br J Sports Med. 2025 Jun 3;59(12):866-876. doi: 10.1136/bjsports-2024-108589. PMID 40049759
- [Result] Olivo G, Nilsson J, Garzon B, Lebedev A, Wahlin A, Tarassova O, Ekblom M, Lovden M. Immediate effects of a single session of physical exercise on cognition and cerebral blood flow: A randomized controlled study of older adults. Neuroimage. 2021 Jan 15;225:117500. doi: 10.1016/j.neuroimage.2020.117500. Epub 2020 Oct 24. PMID 33169699
- [Result] Yildirim MS, Guclu-Gunduz A, Ozkul C, Korkmaz S. Investigating the acute effect of low and moderate intensity aerobic exercise on whole-body task learning and cognition in young adults. Eur J Neurosci. 2024 Sep;60(6):5203-5216. doi: 10.1111/ejn.16504. Epub 2024 Aug 13. PMID 39136270
- [Result] Basso JC, Suzuki WA. The Effects of Acute Exercise on Mood, Cognition, Neurophysiology, and Neurochemical Pathways: A Review. Brain Plast. 2017 Mar 28;2(2):127-152. doi: 10.3233/BPL-160040. PMID 29765853